CLINICAL TRIAL: NCT02499809
Title: The Effects of Vibration Therapy as a Recovery Tool After Intense Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wingate Institute (Other)
Responsible Party: Principal Investigator, Dr. Eyal Shargal, Director, Wingate Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Tarntula 1
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Recovery Method; Muscle Performance; Vibration Therapy
Keywords: Vibration therapy; Recovery from exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Passive (Experimental): Passive recovery
  Interventions: Other: Recovery mode
- Vibration (Experimental): Vibration recovery
  Interventions: Other: Recovery mode

INTERVENTIONS:
Other: Recovery mode — After the gradual maximal exercise the subjects will use different recovery modes (vibration therapy or passive and active recovery).

SUMMARY:
High intensity exercise can lead to muscle damage, resulting in muscle soreness, swelling and reduction in muscle strength. If the recovery is not sufficient or efficient it can increase the risk for injury and decrease the ability of the athlete to perform repetitive exercise and maintain overall performance.

There are a variety of recovery aids which are being used by athletes, such as: the use of compression garments, massage, cold water immersion, sauna etc. Additional recovery strategy currently growing in popularity is the application of vibration.

The evidences regarding the benefits of vibration therapy as a recovery aid are limited, specifically in athlete. Therefore, the proposed study will examine the use of vibration therapy as a recovery tool. The efficacy of this technique will be measure using functional and field tests.

DETAILED DESCRIPTION:
Introduction High intensity exercise can lead to muscle damage, resulting in muscle soreness, swelling and reduction in muscle strength (Proske & Allen, 2005). If the recovery is not sufficient or efficient it can increase the risk for injury and decrease the ability of the athlete to perform repetitive exercise and maintain overall performance. Therefore, the use of recovery strategies between practice sessions can be an important factor in the training process, and will allow the athlete to make the most out of the training regime he or she perform.

There are a variety of recovery aids which are being used by athletes, such as: the use of compression garments, massage, cold water immersion, sauna etc. Additional recovery strategy currently growing in popularity is the application of vibration (Rhea et al. 2009; Broadbent et al. 2010). It has been suggested that the application of vibration could increase the blood flow to the muscle, increase muscle temperature, increases metabolite removal rate and accelerate muscle tissue remodeling. All these processes could reduce delayed onset muscle soreness (DOMS) and accelerate muscle recovery (Rhea et al. 2009; Broadbent et al. 2010; Lau et al. 2011).

Although DOMS are one of the symptoms of muscle damage, they don't necessarily reflect or provide indication of the ability of the muscle to produce strength. That is, it is possible that an athlete will feel well (with no associated pain) but the ability to produce force is still low compare to baseline measurements.

The ability to produce force is an objective and important measure to quantify the recovery status of an athlete after intense exertion (Warren et al. 1999). The efficacy of vibration therapy for promoting recovery has been tested on a small number of studies with equivocal results. For example, Barnes et al. (2012) tested 8 healthy males who completed 300 eccentric contractions of the quadriceps of one leg on an isokinetic dynamometer. Immediately after exercise and 12 and 24 hours post-exercise, the subjects underwent either vibration therapy or a control treatment - no use of any recovery technique. The vibration therapy included 5 sets of 1min vibration at 26 Hz, with 6 mm peak-to-peak displacement. After two weeks after the initial trial, the subjects completed the second trial using the contralateral leg and other treatment. The study's results revealed that the use of vibration therapy reduced muscle peak force and average peak force 24 hours after the eccentric exercise compared to the control group. Another study tested the use of vibration therapy on muscle recovery and strength. This study found that the recovery of elbow flexor peak isometric torque was unaffected by vibration in untrained participants (Lau et al. 2010). This was further supported by Fuller et al. (2014), who found the use of vibration therapy didn't have an additional contribution to recovery after intense exercise compared to stretching or massage.

The evidences regarding the benefits of vibration therapy as a recovery aid are limited. From the paucity of studies in this area it is suggested that there are no additional benefits for using vibration therapy. Yet, the use of different vibration techniques is currently quite popular among athletes and the several studies performed until today were done on non-athlete populations. Furthermore, these studies haven't tested functional variables such as the ability to produce power and performed a repeated performance. Performing a repeated exercise is similar to situations occasionally occur during ball games. Therefore, the proposed study will examine the use of vibration therapy as a recovery tool. The efficacy of this technique will be measure using functional and field tests.

Study purpose The purpose of the proposed study is to examine the effect of vibration therapy as a recovery tool on the ability to perform repeated exertion.

Method The study and its procedures will receive ethic approval by the Helsinki board at Hillel Yaffe Medical Center, Hadera, Israel. The proposed study sample will include 30 novice athletes (18-35 yrs.), who will be recruited to participate in this study.

Inclusion criteria for all groups: (a) participation in physical activity up to three hours per week presently and in the previous year, (b) healthy individuals.

Exclusion criteria for all groups: (a) chronic diseases (hypertension, diabetes, etc.) (b) chronic/frequent use of medications, (c) orthopedic or neurologic injury or disorder.

Exclusion criteria from the study: development of associated muscle or skeletal pain.

Study protocol The participants will arrive at the Ribstein Center for Sports Medicine and Research at the Wingate Institute on two different occasions, 7 days apart.

First visit - a gradual stress test will be performed until exhaustion. Immediately at the end of the test a ten minute recovery period will take place, in which either recovery methods will be used (passive and active or vibration technique). Immediately following the recovery period the participants will perform two functional tests to examine their muscle power and endurance. The 1st test will be countermovement jump (3 jumps will be performed with 15sec rest in between). The 2nd test will be 30sec jump test (continuous jumps). Two minutes resting period will be taken between the tests. The tests will be performed using the Optojump Next measuring system (Optojump, Microgate, Italy).

The recovery methods are:

1. Active and passive: 3min slow walking (4 km/h), 2min standing, 5min slow walking (4 km/h).
2. Vibration therapy: 3min slow walking (4 km/h), 2min standing, 5min vibration therapy with special vibration machine designed for the lower extremities.

At the end of the exercise a peripheral blood sample will be taken from the finger in order to measure blood lactate levels. Additional five samples will be taken in 2min intervals until the end of the recovery period (total of 10min).

Technical information of the vibration machine- vibration frequency between 1-10 hertz, amplitude: 30mm.

Second visit - a gradual stress test will be performed until exhaustion. Immediately at the end of the test a ten minute recovery period will take place, in which the other recovery method will be used (passive and active or vibration technique). Afterwards the two functional tests will be performed.

** The order of the recovery methods will be assigned randomly between the participants.

First visit protocol:

1. Explanation and consent form sign
2. Filling medical questionnaire
3. Medical interview and examination by a sport's physician
4. Anthropometric measures: height, weight, percentage body fat
5. Stress test - including ECG and blood pressure monitoring
6. Recovery - 10min - use of different recovery mode
7. Countermovement jumps test and 30sec jump test Second visit protocol: (7 days apart)

1. Stress test 2. Recovery - 10min - using the other recovery mode not being used at the first visit 3. Countermovement jumps test and 30sec jump test

Measures to be taken during the study:

1. Lactate levels
2. Heart rate (will be monitor continuously during the exercise and during the recovery period)
3. Rate of perceived exertion - subjective evaluation of the difficulty level of the exercise (during the exercise, at the end and after the jumps' tests)
4. Jumps' height during the test, consistency and fatigue index Statistical analysis Paired t-tests will be performed in order to evaluate the effects of the recovery modes on muscle fatigue index and muscle performance measures (power, jump height, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the study
* Active athletes who exercise at least 3 times per week and not less than 3 weekly hours
* Healthy - no chronic disease or orthopedic and neurological disorder
* Not taking any medications on a daily basis

Exclusion Criteria:

* Sedentary
* Medical condition that can affect muscle function

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Muscle performance | 5 minutes
  The height countermovement jump and 30 seconds jump test will be measured after the 10min recovery period.

SECONDARY OUTCOMES:
Blood lactate removal | Straight after the end of the exercise and 5 samples every 2min for an overall of 10min
Rate of perceived exertion | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shargal, PhD, Study Director — Wingate Institute
Locations (1):
- Wingate Institute, Netanya, Israel